CLINICAL TRIAL: NCT02117856
Title: A Randomized Clinical Trial Comparing Patient Satisfaction and Prosthetic Outcomes With Mandibular Implant Overdentures Retained by 1 or 2 Implants
Brief Title: Complete Lower Dentures on 1 or 2 Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Straumann Canada Ltd. (Unknown)
Responsible Party: Principal Investigator, Ross Bryant, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H02-70082
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Tooth-loss; Edentulous Mouth; Complete Denture; Complete Lower Denture
Keywords: Implant-Supported Denture; Single-Implant Denture; Patient Satisfaction; Edentulous Mandible; Dental Implants; Standard of Care; Randomized Clinical Trial
MeSH Terms: conditions — Anodontia; Mouth, Edentulous; Patient Satisfaction | interventions — Coe Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 implant (Active Comparator): Participants receive the following:
  1 implant placed surgically in the mandibular midline; Soft reline of the existing complete lower denture; 2.25mm ball patrix placed on 1 healed implant; and Reline with 1 retentive matrix in the lower denture.
  Interventions: Procedure: 1 implant placed surgically in the mandibular midline; Procedure: Soft reline (Coe Comfort) of the existing complete lower denture; Device: 2.25mm ball patrix placed on 1 healed implant; Procedure: Reline (Ivoclar acrylic-resin) with 1 retentive matrix in the lower denture
- 2 implants (Active Comparator): Participants receive the following:
  2 implants placed surgically in the mandibular canine sites; Soft reline of the existing complete lower denture; 2.25mm ball patrices placed on 2 healed implants; and Reline with 2 retentive matrices in the lower denture.
  Interventions: Procedure: 2 implants placed surgically in the mandibular canine sites; Procedure: Soft reline (Coe Comfort) of the existing complete lower denture; Device: 2.25mm ball patrices placed on 2 healed implants; Procedure: Reline (Ivoclar acrylic-resin) with 2 retentive matrices in the lower denture

INTERVENTIONS:
Procedure: 1 implant placed surgically in the mandibular midline — Participants receive an implant in the mandibular midline using a surgical flap procedure with local anaesthesia.
  Other Names: Implant is Solid Screw, SLA surface, Straumann Canada
  Arms: 1 implant
Procedure: 2 implants placed surgically in the mandibular canine sites — Participants receive implants bilaterally in the site of the mandibular canines using a surgical flap procedure with local anaesthesia.
  Other Names: Implants are Solid Screw, SLA surface, Straumann Canada
  Arms: 2 implants
Procedure: Soft reline (Coe Comfort) of the existing complete lower denture — Participants receive a soft reline of the existing complete lower denture approximately 10 days after placement of the implant(s).
  Other Names: Soft reline is Coe Comfort, GC Corporation
Device: 2.25mm ball patrix placed on 1 healed implant — A 2.25mm ball patrix is screwed onto the 1 implant approximately six weeks after placement of the implant.
  Other Names: Patrix is Spherical Stud Retentive Anchor, Straumann Canada
  Arms: 1 implant
Device: 2.25mm ball patrices placed on 2 healed implants — 2.25mm ball patrices are screwed onto the 2 implants approximately six weeks after placement of the implants.
  Other Names: Patrix is Spherical Stud Retentive Anchor, Straumann Canada
  Arms: 2 implants
Procedure: Reline (Ivoclar acrylic-resin) with 1 retentive matrix in the lower denture — Participants have their complete lower denture relined with a laboratory-processed acrylic resin to incorporate 1 retentive matrix in the denture-base to retain on the implant.
  Other Names: Reline is Ivoclar acrylic-resin, Ivoclar Vivaent Inc, Canada; Matrix is Straumann Gold Matrix, Straumann Canada
  Arms: 1 implant
Procedure: Reline (Ivoclar acrylic-resin) with 2 retentive matrices in the lower denture — Participants have their complete lower denture relined with a laboratory-processed acrylic resin to incorporate 2 retentive matrices in the denture-base to retain on the implants
  Other Names: Reline is Ivoclar acrylic-resin, Ivoclar Vivaent Inc, Canada; Matrix is Straumann Gold Matrix, Straumann Canada
  Arms: 2 implants

SUMMARY:
This study is a randomized clinical trial to compare patient satisfaction and prosthetic outcomes with lower dentures retained by one or two implants. The investigators long-term objective is to establish evidence of the cost-effectiveness of a single implant intervention for improving tolerance to complete dentures. The investigators MAIN AIM will be to investigate patient satisfaction between and within groups with mandibular dentures retained by one or two implants over five years, and SECONDARILY to investigate the survival of implants, and the frequency of events to maintain the dentures and prosthetic attachments as clinically serviceable. Furthermore, multivariate analysis can assess the prediction of patient satisfaction with implant dentures based on various possible factors including age, health, demography and socioeconomic status, number of implants, and maintenance needs. Patient satisfaction will be measured by means of Visual Analogue Scales (VAS) including a measure of overall satisfaction and various specific aspects of satisfaction such as appearance, stability and comfort of the dentures.

The CENTRAL HYPOTHESIS is that mandibular complete dentures retained by single implants are at least as satisfying to patients over a five years period as those retained by two implants for the same period.

The SECONDARY HYPOTHESES are that:

i) there is no difference over five years between groups in the survival of original implants, or in the number of events for maintenance of the dentures or implant attachments; and ii) using each treatment group as it's own control, there is no change in patient satisfaction with lower dentures retained by either one or two implants during the five year loading period.

ELIGIBILITY:
Inclusion Criteria:

* functional in English or accompanied by a responsible adult who can provide translation services
* able to consent to, and participate in, the treatment provided
* available for the duration of the study
* edentulous and with at least six month's experience with conventional complete dentures
* currently wearing conventional complete dentures that are esthetically satisfactory to the patient and technically acceptable in the judgment of the study prosthodontist(s)
* medically/psychologically suitable for implant surgery in the judgment of the study dentists

Exclusion Criteria:

* insufficient alveolar bone height for implant(s) (< 10 mm)
* history of head and neck radiation
* systemic or neurological disease, including: American Society of Anesthesiologists (ASA) Class 3 with recently diagnosed severe systemic disease, e.g. recent (within 6 months) myocardial infarction or stroke; risks associated with bacteraemia, e.g. immune compromise, steroids, in-dwelling catheters, stents, prosthetic heart valves, etc.; Type 1 diabetes, pituitary and adrenal insufficiency, and untreated hypothyroidism; chronic granulomatous disease, e.g. tuberculosis and sarcoidosis; bone disease, e.g. histiocytosis X, Paget's disease, fibrous dysplasia; history of congenital or acquired uncontrolled bleeding, e.g. coumadin
* previous oral implant treatment
* need for additional pre-prosthetic surgery
* need for new complete dentures
* medically/psychologically unsuitable for surgery in the opinion of the study dentists

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2002-11; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Self-assessed VAS satisfaction with the mandibular denture | Annually during 10 years after attaching the mandibular implant denture
  Self-assessed satisfaction is measured on a 10 cm uninterrupted visual analogue scale (VAS) representing a continuum of feelings, with "unsatisfied" at one end and "satisfied" at the other. Each participant makes a global assessment of their satisfaction by marking an X on the line at a point corresponding to their response to the question: "How would you evaluate your 'overall satisfaction' with your lower denture?". A research assistant translates the mark into a number from 0 to 100 by superimposing a template with numbered intervals from 0 to 100 mm.

SECONDARY OUTCOMES:
Change in self-assessed VAS satisfaction with the mandibular denture | From baseline (before implants) to each annual followup for 10 years after attaching the mandibular implant denture
  Self-assessed satisfaction is measured on a 10 cm uninterrupted visual analogue scale (VAS) representing a continuum of feelings, with "unsatisfied" at one end and "satisfied" at the other. Each participant makes a global assessment of their satisfaction by marking an X on the line at a point corresponding to their response to the question: "How would you evaluate your 'overall satisfaction' with your lower denture?". A research assistant translates the mark into a number from 0 to 100 by superimposing a template with numbered intervals from 0 to 100 mm.
Cumulative Implant Survival | During the 10 years after attaching the mandibular implant denture
  Cumulative implant survival was judged by the time to the presence of clinical mobility, pain or suppuration associated with the original mandibular implants.
The frequency of prosthetic maintenance events for the mandibular implant overdenture | During 10 years after attaching the mandibular implant denture
  The frequency of prosthetic maintenance treatment events for the mandibular denture including adjustment, reattachment, or replacement of implant attachment components, and denture base fractures, relining or rebasing, and denture replacement with a new lower denture.
Time to provide the initial surgical and prosthetic treatment for the mandibular implant overdenture intervention | From baseline (before implants) until attachment of the mandibular implant denture, 6 weeks after implant placement
  This is the total professional chair-time recorded to provide the initial surgical and prosthetic treatment for the mandibular implant overdenture intervention.
Costs to provide the initial surgical and prosthetic treatment for the mandibular implant overdenture intervention | From baseline (before implants) until attachment of the mandibular implant denture, 6 weeks after implant placement
  This is the total cost of components and professional and dental laboratory fees to provide the initial surgical and prosthetic treatment for the mandibular implant overdenture intervention.
Time to provide prosthetic maintenance treatment for the mandibular implant overdenture | During 1 year after attachment of the mandibular implant denture
  This is the total professional chair-time recorded to provide prosthetic maintenance treatment for the maxillary denture and the mandibular implant overdenture including contour adjustments, and adjustment, reattachment, or replacement of implant attachment components, and denture repairs, relining or rebasing.
Costs to provide prosthetic maintenance treatment for the mandibular implant overdenture | During 1 year after attachment of the mandibular implant denture
  This is the total cost of components and professional and dental laboratory fees to provide prosthetic maintenance treatment for the maxillary denture and the mandibular implant overdenture including contour adjustments, and adjustment, reattachment, or replacement of implant attachment components, and denture repairs, relining or rebasing.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Bryant, DDS, PhD, Principal Investigator — University of British Columbia; Michael I. MacEntee, LDS, PhD, Study Director — University of British Columbia; Joanne N. Walton, DDS, Study Director — University of British Columbia
Locations (1):
- Department of Oral Health Sciences, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Walton JN, MacEntee MI. Choosing or refusing oral implants: a prospective study of edentulous volunteers for a clinical trial. Int J Prosthodont. 2005 Nov-Dec;18(6):483-8. PMID 16335167
- [Background] Walton JN, MacEntee MI. Screening and enrolling subjects in a randomized clinical trial involving implant dentures. Int J Prosthodont. 2008 May-Jun;21(3):210-4. PMID 18548957
- [Result] Walton JN, Glick N, Macentee MI. A randomized clinical trial comparing patient satisfaction and prosthetic outcomes with mandibular overdentures retained by one or two implants. Int J Prosthodont. 2009 Jul-Aug;22(4):331-9. PMID 19639067
- [Result] Gonda T, Maeda Y, Walton JN, MacEntee MI. Fracture incidence in mandibular overdentures retained by one or two implants. J Prosthet Dent. 2010 Mar;103(3):178-81. doi: 10.1016/S0022-3913(10)60026-1. PMID 20188240
- [Result] Bryant SR, Walton JN, MacEntee MI. A 5-year randomized trial to compare 1 or 2 implants for implant overdentures. J Dent Res. 2015 Jan;94(1):36-43. doi: 10.1177/0022034514554224. Epub 2014 Oct 27. PMID 25348544